Effects of Two Psychosocial Wellness Workshops on Sleep, Stress Management and Wellbeing: Exploration of Psychophysiological Mechanisms

**Brief title:** Student Wellness Workshop study (SWW)

NTC number: not yet assigned

**Date of document:** 12/15/2017

Student Wellness Workshop study (SWW) Statistical Analysis Plan

Statistical analysis will be conducted in IBM SPSS 24.0 using Linear Mixed Models and selective post-hoc comparisons focusing on within-group change for YESplus and WOW at post and follow-up compared to pre-workshop. For each model, results will be reported for main effects of Visit (pre, post, follow-up) and Group (YESplus, WOW), as well as Visit x Group interaction. However, due to limited statistical power of this sample to detect interactions, analysis will focus on within-group change from pre- to post-workshop, as well as pre to follow-up, and corresponding within-group effect size. Thus, to balance type I and type II error with these within-group comparisons, a Bonferroni correction will be applied by multiplying uncorrected *p* values by 4 (the number of post-hoc comparisons per model), allowing alpha to remain at .05 for significance. Effect size estimates will be calculated with Cohen's *d*.